CLINICAL TRIAL: NCT00309946
Title: Phase II Study of AZD2171 (NSC#732208) in Patients With Malignant Mesothelioma
Brief Title: Cediranib Maleate in Treating Patients With Malignant Mesothelioma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00126; N01CM17102 (NIH); CDR0000463521 (Registry Identifier: PDQ (Physician Data Query)); 14203B
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Results first posted 2013-09-10 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2013-10

CONDITIONS: Advanced Malignant Mesothelioma; Epithelial Mesothelioma; Localized Malignant Mesothelioma; Recurrent Malignant Mesothelioma; Sarcomatous Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Initial cediranib maleate dosing was 45 mg (once daily) during a 28-day cycle. Courses repeated every 28 days in the absence of disease progression or unacceptable toxicity. Due to substantial toxicity, the starting dose was subsequently lowered to 30 mg daily.
  Interventions: Drug: cediranib maleate

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin

SUMMARY:
This phase II trial is studying how well cediranib maleate works in treating patients with malignant mesothelioma that cannot be removed by surgery. Cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor

DETAILED DESCRIPTION:
We conducted a multi-center phase II trial of cediranib in patients with unresectable, histologically-confirmed malignant mesothelioma (MM) who had received <=1 prior regimen of chemotherapy. The primary endpoint was objective response rate. Initial cediranib dosing was 45 mg daily during a 28-day cycle. Due to substantial toxicity, the starting dose was subsequently lowered to 30 mg daily.

Pretreatment evaluation included a medical history and physical exam, complete blood count and differential, chemistry panel, pregnancy test, and a computed tomography (CT) scan of the chest, abdomen, and pelvis if relevant. A history and physical exam were repeated every 14 days and laboratory evaluations including a complete blood count with differential, serum chemistry panel, and urinalysis were repeated every 7 days. Patients were provided with a blood pressure monitoring device and a diary to record their blood pressure readings twice daily.

Patients received a minimum of 2 cycles unless unacceptable toxicity or rapid clinical progression of disease occurred. Response was evaluated by CT imaging every two cycles. Confirmatory scans were to be obtained at least 4 weeks after initial documentation of an objective complete or partial response.

Cediranib was administered orally once daily on days 1 through 28 of a 28-day cycle. Cediranib was initially dosed at 45 mg daily, but due to substantial rates of toxicity the protocol was amended in June 2007 to decrease the starting dose to 30 mg daily. Cediranib was taken 1 hour (h) before or 2 h after meals. Only one dose modification was permitted. When the starting cediranib dose was 45 mg, dose level-1 was 30 mg daily. After the protocol amendment, dose level-1 was 20 mg daily. Further dose reductions were allowed at the discretion of the investigator only if the patient had received clinical benefit from cediranib for >3 months. Patients undergo blood collection periodically during study for biomarker and optional pharmacogenomic correlative studies. After completion of study treatment, patients are followed for up to 8 weeks.

Adverse effects were graded according to National Cancer Institute Common Toxicity Criteria version 3.0. The dose was reduced for grade 3 or greater non-hematologic toxicity attributable to cediranib or grade 4 hematologic toxicity if the toxicity lasted for >5 days and did not resolve to <=grade 2. Maximal antihypertensive therapy was defined as taking 4 antihypertensive agents for >2 weeks at full dosage. For patients on antihypertensive therapy who had an elevation in systolic blood pressure (SBP) >=140 mmHg or diastolic blood pressure (DBP) >=90 mmHg on 2 separate readings during a 48 h period, the dose of cediranib was maintained without interruption while the dosage of current antihypertensive therapy was increased or an additional antihypertensive agent was started. If 2 readings reported a SBP >=180 mmHg or a DBP >=105 mmHg during a 1 week period, cediranib was held and there was either an increase in the dosage of current antihypertensive therapy or an additional antihypertensive agent was added. Resumption of cediranib was allowed only after the blood pressure was <140/90 mmHg. If 2 blood pressure readings recorded an SBP >=160 mmHg or a DBP >=105 mmHg 1 h apart during a 48 hour period in a patient already on maximal antihypertensive therapy, cediranib was held and treatment was resumed at 1 dose level lower when the blood pressure was <160/105.

PRIMARY OBJECTIVE:

I. Determine the objective response rate in patients with malignant pleural, peritoneal, or tunica vaginalis mesothelioma that is not amenable to curative surgery who are treated with AZD2171 (cediranib maleate).

SECONDARY OBJECTIVES:

I. Determine the progression-free survival of patients treated with AZD2171. II. Determine the toxicity experienced by patients treated with AZD2171. III. Determine median and overall survival of patients treated with AZD2171.

TERTIARY OBJECTIVES:

I. Generate preliminary data regarding potential utility of pharmacogenomic and plasma/serum biomarkers of angiogenesis as predictive or prognostic markers for future investigations of this drug in malignant mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed malignant pleural, peritoneal, or tunica vaginalis mesothelioma

  * Epithelial, sarcomatoid, or mixed subtype
* International Mesothelioma Interest Group stage II-IV disease (for patients with pleural mesothelioma)
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR > 10 mm by spiral CT scan

  * Pleural effusion and ascites are not considered measurable lesions
* Disease not amenable to curative surgery
* No known brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 OR Karnofsky PS 70-100%
* Life expectancy > 3 months
* White blood cell (WBC) ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin ≥ 8 g/dL
* Platelets ≥ 100,000/mm³
* Total bilirubin normal
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal(ULN)
* Creatinine normal OR creatinine clearance > 60 mL/min
* Fertile patients must use effective contraception
* Not pregnant or nursing
* Negative pregnancy test
* No history of allergic reactions to compounds of similar chemical or biologic composition to AZD2171
* Mean corrected QT interval (QTc) ≤ 500 msec (with Bazett's correction) by EKG
* No history of long QT syndrome
* Proteinuria ≤ 1+ on two consecutive dipsticks taken ≥ 1 week apart
* No other concurrent malignancy
* No New York Heart Association class III or IV cardiac disease
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Hypertension
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situations that would limit study compliance
* No more than 1 prior cytotoxic chemotherapy

  * Prior intrapleural cytotoxic agents (including bleomycin) do not count towards prior cytotoxic chemotherapy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* No prior radiotherapy to the only site of measurable disease
* At least 4 weeks since prior radiotherapy and recovered
* At least 4 weeks since prior major surgery and recovered
* More than 30 days since prior participation in an investigational trial
* No prior treatment with a vascular endothelial growth factor (VEGF) inhibitor
* No other concurrent investigational agents
* No concurrent commercial agents for the malignancy
* No concurrent medication that may markedly affect renal function (e.g., vancomycin, amphotericin, or pentamidine)
* No concurrent hematopoietic growth factors except epoetin alfa
* No concurrent palliative radiotherapy
* No combination antiretroviral therapy for HIV-positive patients
* No concurrent drugs or biologics with proarrhythmic potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hedy Kindler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Campbell NP, Kunnavakkam R, Leighl N, Vincent MD, Gandara DR, Koczywas M, Gitlitz BJ, Agamah E, Thomas SP, Stadler WM, Vokes EE, Kindler HL. Cediranib in patients with malignant mesothelioma: a phase II trial of the University of Chicago Phase II Consortium. Lung Cancer. 2012 Oct;78(1):76-80. doi: 10.1016/j.lungcan.2012.06.011. Epub 2012 Jul 23. PMID 22831987

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 51
Completed | 50
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 64 [44 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate, Complete (CR) or Partial (PR) Response
Description: Evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. To be assigned a status of PR or CR, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 4 weeks after the criteria for response are first met.
Time Frame: Every 8 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 50
percentage of participants | 5

2. Secondary Outcome: Changes in Laboratory Correlates
Description: Examined using paired t-test or Wilcoxon signed-ranks test.
Time Frame: Baseline, days 15 and 29 of course 1, and then every 28 days
Population: This outcome was not measured/assessed for any of the study subjects.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Pharmacogenomics by Correlating Genetic Polymorphisms With Drug Activity and Toxicity
Description: Focus on variants of genes in the pathway targeted by cediranib maleate, including kdr/flk-1 (the specific target of cediranib maleate) and the genes that encode Vascular endothelial growth factor A (VEGF-A) or HIF1α. If additional information relevant to other genes of interest in the pathway becomes available the samples will be utilized for such analysis as well.
Time Frame: Week 1 of course 1
Population: This outcome was not measured/assessed for any of the study subjects.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: After completion of study treatment, patients are followed for up to 8 weeks.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 31/51
Other Adverse Events (participants affected / at risk) | 49/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=51)
Abdominal distension (Gastrointestinal disorders) | 1 — Abdominal distension occurs when substances, such as air (gas) or fluid, accumulate in the abdomen causing its outward expansion beyond the normal girth of the stomach and waist.
Abdominal pain (General disorders) | 1 — Pain in the abdominal region
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 — Increased levels of alanine aminotransferase, indicative of liver damage or disease.
Anaphylaxis (Immune system disorders) | 1 — Anaphylaxis is a serious allergic reaction that is rapid in onset and may cause death.
Anorexia (Gastrointestinal disorders) | 1 — Anorexia is the decreased sensation of appetite.
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 1 — Increased levels of aspartate aminotransferase (AST)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 — Atelectasis is defined as the collapse or closure of the lung resulting in reduced or absent gas exchange.
Atrial flutter (Cardiac disorders) | 1 — Atrial flutter (AFL) is an abnormal heart rhythm that occurs in the atria of the heart.
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 — Bronchopulmonary hemorrhage is a disorder characterized by bleeding from the bronchial wall and/or lung parenchyma.
Cardiac arrest (Cardiac disorders) | 1 — Cardiac arrest, also known as cardiopulmonary arrest or circulatory arrest, is the cessation of normal circulation of the blood due to failure of the heart to contract effectively.
Chest wall pain (General disorders) | 3 — Pain in the chest wall not attributed to any cardiac disorder.
Cognitive disturbance (Nervous system disorders) | 1 — A disorder characterized by a conspicuous change in cognitive function.
Conduction disorder (Cardiac disorders) | 1 — Impairment of conduction in heart excitation; often applied specifically to atrioventricular heart block.
Confusion (Nervous system disorders) | 2 — Loss of orientation (ability to place oneself correctly in the world by time, location, and/or personal identity sometimes accompanied by disordered consciousness and often memory (ability to correctly recall previous events or learn new material).
Constipation (Gastrointestinal disorders) | 2 — Constipation (also known as costiveness or dyschezia) refers to bowel movements that are infrequent or hard to pass.
Creatinine increased (Metabolism and nutrition disorders) | 1 — Increased levels of creatinine
Dehydration (Gastrointestinal disorders) | 2 — Dehydration is the excessive loss of body water
Depressed level of consciousness (Nervous system disorders) | 1 — A neurologic state characterized by decreased ability to perceive and respond.
Diarrhea (Gastrointestinal disorders) | 2 — Condition of having three or more loose or liquid bowel movements per day
Dizziness (Nervous system disorders) | 1 — Dizziness is an impairment in spatial perception and stability.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 — Dyspnea - shortness of breath.
ECG QTc interval prolonged (Cardiac disorders) | 1 — Electrocardiogram QT corrected interval prolonged
Encephalopathy (Nervous system disorders) | 1 — Syndrome of global brain dysfunction
Failure to thrive (General disorders) | 1 — Insufficient weight gain or inappropriate weight loss.
Fatigue (General disorders) | 2 — Fatigue (also called exhaustion, tiredness, lethargy, languidness, languor, lassitude, and listlessness) is a subjective feeling of tiredness which is distinct from weakness, and has a gradual onset.
Headache (General disorders) | 1 — Pain in the head or neck region.
Hyperglycemia (Metabolism and nutrition disorders) | 1 — Hyperglycemia, or high blood sugar is a condition in which an excessive amount of glucose circulates in the blood plasma.
Hyperkalemia (Metabolism and nutrition disorders) | 1 — Hyperkalemia refers to the condition in which the concentration of the electrolyte potassium in the blood is elevated.
Hypertension (Cardiac disorders) | 4 — Elevated blood pressure in the arteries
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 — Hypoalbuminemia is a medical condition where levels of albumin in blood serum are abnormally low.
Hypoglycemia (Metabolism and nutrition disorders) | 1 — Hypoglycemia is an abnormally diminished content of glucose in the blood.
Hyponatremia (Metabolism and nutrition disorders) | 1 — Hyponatremia - An electrolyte disturbance in which the sodium ion concentration in the serum is lower than normal.
Hypotension (Cardiac disorders) | 1 — Hypotension is low blood pressure.
Infection with unknown ANC: Blood (Infections and infestations) | 1 — Blood infection with unknown Absolute Neutrophil Count (ANC)
Intracranial hemorrhage (General disorders) | 1 — An intracranial hemorrhage (ICH) is a hemorrhage, or bleeding, within the skull.
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 — Infection in the lung
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 — Lymphocyte count decreased
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 — Second-degree atrioventricular (AV) block is a disease of the electrical conduction system of the heart. It refers to a conduction block between the atria and ventricles.
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 — Muscle weakness or myasthenia is a lack of muscle strength.
Pericardial effusion (Cardiac disorders) | 1 — Pericardial effusion ("fluid around the heart") is an abnormal accumulation of fluid in the pericardial cavity.
Peripheral motor neuropathy (Nervous system disorders) | 1 — A disorder characterized by inflammation or degeneration of the peripheral motor nerves.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 — Pleural effusion is excess fluid that accumulates between the two pleural layers, the fluid-filled space that surrounds the lungs.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 — A pneumothorax is an abnormal collection of air or gas in the pleural space that separates the lung from the chest wall and which may interfere with normal breathing.
Proteinuria (Renal and urinary disorders) | 2 — Proteinuria-also called albuminuria or urine albumin-is a condition in which urine contains an abnormal amount of protein
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 — Pulmonary embolism (PE) is a blockage of the main artery of the lung or one of its branches by a substance that has traveled from elsewhere in the body through the bloodstream (embolism).
Seizure (Nervous system disorders) | 2 — A seizure is the physical findings or changes in behavior that occur after an episode of abnormal electrical activity in the brain.
Sepsis (Infections and infestations) | 1 — Sepsis is a potentially deadly medical condition characterized by a whole-body inflammatory state (called a systemic inflammatory response syndrome or SIRS) caused by severe infection.
Sinus tachycardia (Cardiac disorders) | 1 — Sinus tachycardia is a heart rhythm with elevated rate of impulses originating from the sinoatrial node, defined as a rate greater than 100 beats/min (bpm) in an average adult.
Small intestinal obstruction (Gastrointestinal disorders) | 1 — Intestinal obstruction is a blockage that keeps food or liquid from passing through the small intestine.
Thromboembolic event (Vascular disorders) | 4 — Formation of a blood clot inside a blood vessel, obstructing the flow of blood through the circulatory system.
Urinary retention (Renal and urinary disorders) | 1 — Urinary retention is the inability to empty the bladder.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=51)
Abdominal pain (General disorders) | 8 — Pain in the abdominal region.
Alanine aminotransferase (ALT) increased (Metabolism and nutrition disorders) | 11 — Increased levels of alanine aminotransferase, indicative of liver damage or disease.
Alkaline phosphatase (ALP) increased (Metabolism and nutrition disorders) | 9 — Increased levels of Alkaline phosphatase
Allergic rhinitis (Immune system disorders) | 4 — Allergic rhinitis is an allergic inflammation of the nasal airways.
Anemia (Blood and lymphatic system disorders) | 23 — Anemia is a decrease in number of red blood cells (RBCs) or less than the normal quantity of hemoglobin in the blood.
Anorexia (Gastrointestinal disorders) | 28 — Anorexia is the decreased sensation of appetite.
Anxiety (Nervous system disorders) | 5 — Anxiety is an unpleasant state of inner turmoil and apprehension, often accompanied by nervous behavior, such as pacing back and forth, somatic complaints and rumination.
Arthralgia (General disorders) | 4 — Joint pain.
Aspartate aminotransferase (AST) increased (Metabolism and nutrition disorders) | 10 — Increased levels of aspartate aminotransferase (AST)
Back pain (General disorders) | 10 — Pain in the back.
Chest wall pain (General disorders) | 23 — Pain in chest wall
Constipation (Gastrointestinal disorders) | 13 — Constipation (also known as costiveness or dyschezia) refers to bowel movements that are infrequent or hard to pass.
Cough (Respiratory, thoracic and mediastinal disorders) | 12 — A cough is a sudden and often repetitively occurring reflex which helps to clear the large breathing passages from secretions, irritants, foreign particles and microbes.
Creatinine increased (Metabolism and nutrition disorders) | 6 — Increased levels of creatinine
Dehydration (Gastrointestinal disorders) | 3 — Dehydration is the excessive loss of body water
Depression (Nervous system disorders) | 4 — Depression is a mental disorder characterized by episodes of all-encompassing low mood accompanied by low self-esteem and loss of interest or pleasure in normally enjoyable activities.
Diarrhea (Gastrointestinal disorders) | 30 — Diarrhea is the condition of having three or more loose or liquid bowel movements per day.
Dry mouth (Gastrointestinal disorders) | 4 — Dry mouth is associated a change in the composition of saliva or reduced salivary flow (hyposalivation).
Dysgeusia (Gastrointestinal disorders) | 5 — Dysgeusia is a distortion of the sense of taste
Dyspepsia (Gastrointestinal disorders) | 9 — Dyspepsia is a condition of impaired digestion characterized by chronic or recurrent pain in the upper abdomen, upper abdominal fullness and feeling full earlier than expected when eating.
Dysphagia (Gastrointestinal disorders) | 6 — Dysphagia is the medical term for the symptom of difficulty in swallowing.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 — Dyspnea - shortness of breath.
Edema (limb) (Blood and lymphatic system disorders) | 5 — Swelling of tissues in the limbs due to the accumulation of fluids.
Epistaxis (Blood and lymphatic system disorders) | 6 — Nosebleed
Fatigue (General disorders) | 35 — Fatigue (also called exhaustion, tiredness, lethargy, languidness, languor, lassitude, and listlessness) is a subjective feeling of tiredness which is distinct from weakness, and has a gradual onset.
Headache (General disorders) | 9 — Pain in the head or neck region.
Hematuria (Renal and urinary disorders) | 4 — Hematuria is blood in the urine.
Hyperglycemia (Metabolism and nutrition disorders) | 26 — Hyperglycemia, or high blood sugar is a condition in which an excessive amount of glucose circulates in the blood plasma.
Hyperkalemia (Metabolism and nutrition disorders) | 7 — Hyperkalemia refers to the condition in which the concentration of the electrolyte potassium in the blood is elevated.
Hypertension (Cardiac disorders) | 29 — Elevated blood pressure in the arteries.
Hypoalbuminemia (Metabolism and nutrition disorders) | 20 — Hypoalbuminemia is a medical condition where levels of albumin in blood serum are abnormally low.
Hypocalcemia (Metabolism and nutrition disorders) | 4 — Hypocalcemia is the presence of low serum calcium levels in the blood, usually taken as less than 2.1 mmol/L or 9 mg/dl or an ionized calcium level of less than 1.1 mmol/L or 4.5 mg/dL.
Hypoglycemia (Metabolism and nutrition disorders) | 4 — Hypoglycemia is an abnormally diminished content of glucose in the blood.
Hypomagnesemia (Metabolism and nutrition disorders) | 7 — Hypomagnesemia (or hypomagnesaemia) is an electrolyte disturbance in which there is an abnormally low level of magnesium in the blood.
Hyponatremia (Metabolism and nutrition disorders) | 18 — Hyponatremia - An electrolyte disturbance in which the sodium ion concentration in the serum is lower than normal.
Hypotension (Blood and lymphatic system disorders) | 3 — Hypotension is low blood pressure.
Hypothyroidism (Endocrine disorders) | 11 — Hypothyroidism is a state in which the thyroid gland does not produce a sufficient amount of the thyroid hormones thyroxine (T4) and triiodothyronine (T3).
Insomnia (General disorders) | 5 — Insomnia, or sleeplessness, is a sleep disorder in which there is an inability to fall asleep or to stay asleep as long as desired.
Lymphocyte count decreased (Blood and lymphatic system disorders) | 14 — Low lymphocyte count
Mucositis (oral) (Gastrointestinal disorders) | 12 — Inflammation and ulceration that occurs in the mouth
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 — Muscle weakness is a lack of muscle strength.
Nail loss (Skin and subcutaneous tissue disorders) | 4 — Fingernail loss is a removal of the whole or part of the nail from the bed.
Nausea (Gastrointestinal disorders) | 17 — Nausea a sensation of unease and discomfort in the upper stomach with an involuntary urge to vomit.
Oral pain (General disorders) | 4 — Pain in the mouth.
Pain - Other (General disorders) | 6 — Pain in unspecified region.
Pain in extremity (General disorders) | 6 — Pain in extremity
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 — Palmar-plantar erythrodysesthesia (hand-foot) syndrome results when a small amount of drug leaks out of the blood vessels, damaging tissues.
Peripheral sensory neuropathy (Nervous system disorders) | 4 — Inflammation or degeneration of the sensory nerves.
Pharyngolaryngeal pain (Gastrointestinal disorders) | 5 — A disorder characterized by marked discomfort sensation in the pharyngolaryngeal (pharynx/larynx) region.
Platelet count decreased (Blood and lymphatic system disorders) | 8 — Low platelet count
Proteinuria (Renal and urinary disorders) | 14 — Proteinuria-also called albuminuria or urine albumin-is a condition in which urine contains an abnormal amount of protein.
Rash (maculo-papular) (Skin and subcutaneous tissue disorders) | 6 — A maculopapular rash is a type of rash characterized by a flat, red area on the skin that is covered with small confluent bumps.
Sinus tachycardia (Cardiac disorders) | 4 — Sinus tachycardia is a heart rhythm with elevated rate of impulses originating from the sinoatrial node, defined as a rate greater than 100 beats/min (bpm) in an average adult.
Voice changes (Respiratory, thoracic and mediastinal disorders) | 11 — Hoarseness, loss or alteration in voice, laryngitis
Vomiting (Gastrointestinal disorders) | 9 — Vomiting is the forceful expulsion of the contents of one's stomach through the mouth and sometimes the nose.
Weight loss (General disorders) | 12 — Weight loss is a reduction of the total body mass, due to a mean loss of fluid, body fat or adipose tissue and/or lean mass, namely bone mineral deposits, muscle, tendon and other connective tissue.
White blood cell count decreased (Blood and lymphatic system disorders) | 4 — Low white blood cell count

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less